CLINICAL TRIAL: NCT02304497
Title: Evaluation of Platelet Rich Fibrin Growth Factors (PRF) in Type 2 Diabetic Patients With Chronic Periodontitis
Brief Title: PRF Growth Factors Levels in Diabetic Patients With Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Seyma Bozkurt Doğan, PhD, DDS, Bulent Ecevit University
Other Study IDs: 2013-62550515-01
Record Dates: First submitted 2014-11-21; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus; Chronic Periodontitis
Keywords: Diabetes mellitus; Platelet rich fibrin; growth factor
MeSH Terms: conditions — Diabetes Mellitus; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- DM-CTRL: Diabetes mellitus patients with periodontally healthy Platelet Rich Fibrin obtained
  Interventions: Other: Platelet Rich Fibrin
- DM-CP: Diabetes mellitus patients with chronic periodontitis Platelet Rich Fibrin obtained
  Interventions: Other: Platelet Rich Fibrin
- CP: Chronic periodontitis patients with systemically healthy Platelet Rich Fibrin obtained
  Interventions: Other: Platelet Rich Fibrin
- CTRL: Periodontally and systemically healthy subject Platelet Rich Fibrin obtained
  Interventions: Other: Platelet Rich Fibrin

INTERVENTIONS:
Other: Platelet Rich Fibrin — Procedure: Platelet Rich Fibrin obtained

SUMMARY:
Diabetic patients may show different release of growth factors when microvascular complications such as; retinopathy or periodontitis are seen. Diabetes have an adverse effect on periodontal health and periodontal infection have an adverse effect on glycemic control and incidence of diabetes complications. Therefore, the investigators hypothesize that growth factors levels releasing from platelet rich fibrin (PRF) in diabetes mellitus (DM) may be decrease because of periodontitis is considered to be the sixth microvascular complication of diabetes or diabetes may have inductive effect on PRF growth factors levels in periodontal disease. Determination of PRF growth factors levels may be beneficial to treatment of diabetic patient with periodontal disease by using PRF.

DETAILED DESCRIPTION:
The aim of the investigators study was to evaluate levels of platelet derived growth factor-AB (PDGF-AB), vascular endothelial growth factor ( VEGF),transforming growth factor-beta1 and beta 2 (TGF-β1 and β2), basic-Fibroblast growth factor (b-FGF), insulin like growth factor-1 ( IGF-1) in type 2 diabetic (T2DM) patients with chronic periodontitis.

This study consisted of 80 subjects; 20 patients were T2DM with periodontally healthy (DM-CTRL), 20 patients were T2DM with chronic periodontitis (DM-CP ), 20 patients were systemically healthy with chronic periodontitis (CP; ), 20 subjects were systemically and periodontally healthy (CTRL).

Subjects were clinically evaluated with regards to the plaque index (PI), gingival index (GI), probing pockets depth (PD), clinical attachment level (CAL), bleeding on probing (BOP) recorded at six sites per tooth (disto-facial, mid-facial, mesio-facial, mesio-lingual, disto-lingual and mid-lingual) using a periodontal Goldman/Fox Williams probe calibrated in millimeters.

PRF was prepared without biochemical manipulation of blood. Intravenous blood from each patient was collected in 10 ml sterile tubes without anticoagulant by venipuncture of antecubital vein. Immediately test tubes were centrifuged using a centrifugation machine ( Electro.mag M 815 P Laboratory Centrifuge ; Istanbul, Turkey) at 2700 rpm ( approximately 700g ) for 12 min . The centrifuged blood presented with a structured fibrin clot in the middle of the tube just between the red corpuscles at the bottom and acellular plasma at the top. PRF was easily separated from the red corpuscule base using steril scissors and inserted into steril tubes. The tubes were put on a shaker and agitated gently. After 5 minutes, the tubes were vortexed to form a PRF membrane and the volume of releasate was measured and the releasate returned into the tube. The tubes were further agitated gently. Samples were taken at 5th minute and immediately centrifuged at 5000rpm for 15 minutes (Electro.mag M 815 P Laboratory Centrifuge ; Istanbul, Turkey) to pellet any residual blood cells , and were stored at -80 centigrade degree for subsequent assays.

Samples were assayed by using enzyme-linked immunosorbent assay (ELISA) with an ELX 800 G ELISA device (BIO-TEC Instruments, Winooski, USA). The following ELISA kits were used in this study: b-FGF, TGF-β2 and IGF 1 (Assay Biotechnology Company, CA, USA); PDGF-AB, VEGF and TGF-β1 (Boster Biological Technology, CA, USA).

Statistical analysis was performed using a commercially available software (SPSS 15.0; SPSS Inc., Chicago, IL). The Shapiro-Wilk test was used to investigate whether the data were normally distributed. When normal distribution with equal variances was assumed in PDGF-AB, VEGF, TGF-β1, variables were compared using one-way analysis of variance (ANOVA) with Bonferroni post hoc test. If the assumption of normality failed, comparisons of the age, TGF-β2, b-FGF, IGF-1, HbA1c, fasting blood glucose, postprandial blood glucose, full-mouth PD, CAL, GI, PI and BOP were tested using the Kruskal-Wallis non-parametric test followed by post-hoc group comparisons with the Bonferroni-adjusted Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* CP patients required a diagnosis of moderate to advanced CP and showing radiographic evidence of bone loss and, defined as clinical attachment loss with a minimum of 6 teeth having periodontal pocket greater than 4 mm, a minimum of 20 natural teeth,
* No periodontal treatment in the prior 6 months.
* T2DM patients who had HbA1c levels between 6%-8 %
* Periodontally healthy subjects (periodontal pocket depth < 4 mm)

Exclusion Criteria:

* If they had any known systemic diseases other than type 2 diabetes mellitus
* Patient had been under medicine treatment for at least 6 months except patients with diabetes who were treated with stable doses of hypoglycemic agents
* Patients with major complications of DM (i.e., cardiovascular and peripheral vascular diseases
* Insufficient platelet count (<200,000/mm3); 2) pregnancy/lactation )
* Tobacco use
* Pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients participating the study were recruited from indivuduals referred to Department of Periodontology, Faculty of Dentistry, University of Bülent Ecevit University for either dental treatment or dental check-ups.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Platelet Rich Fibrin (PRF) levels of vascular endothelial growth factor (VEGF) | Baseline
PRF levels of platelet derived growth factor- AB (PDGF-AB) | Baseline
PRF levels of basic- fibroblast growth factor (b-FGF) | Baseline
PRF levels of transforming growth factor- beta 1 (TGF-β1) | Baseline
PRF levels of transforming growth factor- beta 2 (TGF-β2) | Baseline
PRF levels of insulin like growth factor -1 (IGF-1) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma Bozkurt Doğan, DDS, Study Chair — Bülent Ecevit University Faculty of Dentistry; Umut Ballı, DDS, Principal Investigator — Bülent Ecevit University Faculty of Dentistry; Figen Öngöz Dede, DDS, Study Director — Bülent Ecevit University Faculty of Dentistry; Mustafa Cenk Durmuşlar, DDS, Principal Investigator — Bülent Ecevit University Faculty of Dentistry; Murat Can, Assoc. Professor, Principal Investigator — Bülent Ecevit University Faculty of Medicine